CLINICAL TRIAL: NCT02149966
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose, Safety, Pharmacokinetic, and Pharmacodynamic Study of Orally Administered AG-348 in Healthy Volunteers
Brief Title: A Phase I Study of AG-348 in Healthy Volunteers
Acronym: AG-348MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG348-C-002
Record Dates: First submitted 2014-05-27; First posted 2014-05-29 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Volunteer
Keywords: safety and tolerability; pharmacokinetic study
MeSH Terms: interventions — mitapivat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AG-348 (Experimental): Multiple oral doses of AG-348
  Interventions: Drug: AG-348
- Placebo (Placebo Comparator): Multiple oral doses of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AG-348 — A range of doses of AG-348 will be tested based on the assessment of safety and tolerability. AG-348 will be administered by mouth (orally) each day for a period of 14 days.
  Arms: AG-348
Drug: Placebo — Placebo will be administered by mouth (orally) each day for a period of 14 days.
  Arms: Placebo

SUMMARY:
This is a dose escalation study that will be conducted in healthy volunteers. Multiple cohorts of volunteers will receive ascending (increasingly higher) oral doses of AG-348 daily for 14 days to evaluate the safety and tolerability of multiple oral doses of AG-348, the pharmacokinetics (PK) of multiple doses of AG-348, and the pharmacodynamic profile of AG-348 with specific biomarkers assessed in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female subjects 18 - 60 years, in good general health who are able to understand consent and complete all study procedures.
* Female subjects of non-child bearing potential (surgically sterile or post-menopausal as confirmed by age [over 50 years], amenorrhea for ≥12 consecutive months and FSH).
* Male subjects who are not vasectomized must agree to use contraception up to 30 days after dosing.
* Subjects with body weight ≥50 kg; BMI ≥18.5 and ≤32 kg/m2.
* Subjects who are non-smokers and have not used nicotine-containing products for at least 3 months prior to screening.
* Subjects must be willing to refrain from caffeine- or xanthene-containing products (coffee, tea, chocolate) for 48 hours prior to dosing through discharge from the clinical facility.
* Subjects must agree to refrain from strenuous exercise starting 72 hours prior to admission through final follow-up visit.
* Subjects must refrain from use of alcohol starting 7 days (14 days for red wine) prior to admission through final follow-up visit.
* Subjects must agree not to donate blood products for duration of study participation.

Exclusion Criteria:

* Subjects who have previously received AG-348.
* Subjects with clinically relevant screening laboratory tests.
* Female subjects who are not post-menopausal.
* Subjects with recent use of prescription, over the counter (OTC), herbal and/or dietary medications and/or supplements.
* Male subjects with QTcF interval ECG > 450 msec,or female subjects with QTcF interval ECG > 470 msec.
* Subjects with a history of a serious mental illness.
* Subjects with a clinically relevant medical history or pre-existing medical condition that would interfere with the absorption, metabolism or excretion of the study drug.
* Subjects with a history of any primary malignancy (cancer). Exceptions are certain skin cancers, cervical cancer in situ or other cancers that have been curatively treated without evidence of disease for a minimum of 1 year.
* Subjects with glucose-6-phosphate-dehydrogenase (G6PD) deficiency.
* Subjects who are positive for hepatitis B, hepatitis C or HIV.
* Subjects who have undergone surgery 6 months prior to screening.
* Subjects who have a history of illicit drug use or alcoholism within the last year.
* Subjects who are participating in other concurrent clinical trial of an investigational drug, or have received another investigational agent within the last 2 months.
* Subjects with any conditions which would make the subject unsuitable for enrollment, or could interfere with the subject's participation in or completion of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 29 days

SECONDARY OUTCOMES:
Pharmacokinetics parameters of AG-348 | 17 days
  Descriptive statistics will be used to summarize PK parameters of AG-348 for each dose group and, where appropriate, for the entire population. Standard non-compartmental PK parameters will be calculated from individual plasma concentration data.
Pharmacodynamic (PD) relationship of AG-348 and metabolic biomarkers | 17 days
  The potential relationship between AG-348 and metabolic biomarkers will be explored with descriptive and graphical methods. Details on the evaluation of pyruvate kinase (PKR) activity and other potential PD biomarkers will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Agresta, MD, MPH & TM, Study Director — Agios Pharmaceuticals, Inc.
Locations (1):
- Baltimore, Maryland, United States

REFERENCES:
- [Derived] Yang H, Merica E, Chen Y, Cohen M, Goldwater R, Kosinski PA, Kung C, Yuan ZJ, Silverman L, Goldwasser M, Silver BA, Agresta S, Barbier AJ. Phase 1 Single- and Multiple-Ascending-Dose Randomized Studies of the Safety, Pharmacokinetics, and Pharmacodynamics of AG-348, a First-in-Class Allosteric Activator of Pyruvate Kinase R, in Healthy Volunteers. Clin Pharmacol Drug Dev. 2019 Feb;8(2):246-259. doi: 10.1002/cpdd.604. Epub 2018 Aug 9. PMID 30091852